CLINICAL TRIAL: NCT05981235
Title: FTiH, Phase 1 Investigator-Initiated Trial (IIT) to Evaluate the Safety, Feasibility, Cellular Kinetics, and Preliminary Antitumor Activity of AZD6422 in Adult Participants With Advanced or Metastatic CLDN18.2+ GI Tumors
Brief Title: Phase 1 Trial of AZD6422 in CLDN18.2+ GI Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9540C00001
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Tumors
Keywords: CLDN18.2+ GI Tumors Solid tumor CAR-T Cell therapy AZD6422
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD6422 (Experimental): It is anti-CLDN18.2 CAR-T cell therapy and the study consists of two parts: dose escalation (part 1) and dose expansion (part 2)
  Interventions: Biological: AZD6422 CLDN18.2 CAR-T product

INTERVENTIONS:
Biological: AZD6422 CLDN18.2 CAR-T product — AZD6422 CAR-T product infusion after pre-conditioning
  Other Names: AZD6422

SUMMARY:
This is a FTiH, Phase 1 IIT to evaluate the safety, feasibility, cellular kinetics (CK), pharmacodynamics (PD), immunogenicity, and preliminary antitumor activity of AZD6422 in adult participants with advanced or metastatic CLDN18.2+ GI tumors.

DETAILED DESCRIPTION:
Qualified researchers can request access to anonymized individual patient-level data from sponsor or the collaborator group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the sponsor disclosure commitment. Yes, indicates that sponsors are accepting requests for IPD, but this does not mean all requests will be shared.

ELIGIBILITY:
Inclusion Criteria:

* 1Capable of giving signed informed consent and keep compliance with the requirements and restrictions listed in the ICF and in this protocol.

  2Age ≥ 18 years at the time of signing the informed consent. 3At least 1 lesion, that qualifies as a RECIST v1.1 target lesion at baseline. Histologically confirmed diagnosis of unresectable or metastatic GI adenocarcinoma that has failed prior lines systemic treatment or with standard anticancer therapy.

  4Confirmation of CLDN18.2 expression determined by IHC . 5ECOG PS of 0 to 1. 6 Life expectancy of > 12 weeks. 7Evidence of appropriate organ function, as determined by clinical laboratory values.

  8Participants of childbearing potential (including woman of childbearing potential and males who have a partner) must take highly effective contraception measure.

Exclusion Criteria:

* 1.Prior treatment with any CAR-T cell therapy. 2.History of upper digestive tract bleeding secondary to previous CLDN18.2-targeting therapies; clinically significant unstable or active peptic ulcer disease or upper digestive tract bleeding 3.Cancer-related spinal cord compression, leptomeningeal disease, or brain metastases.

  4.Receipt of the last dose of anticancer therapy within 5 half-lives or ≤ 21 days prior to apheresis, treatment radiotherapy within 6 weeks (loco-regional palliative radiotherapy within 7 days) prior to apheresis.

  5.Treatment with any anticoagulant or antiplatelet therapy. 6.History of, or active, bleeding diatheses. 7.Active or chronic infection disease (s). 8.History of another primary malignancy ≤ 3 years before enrolment. 9.Any history of autoimmune neurological conditions. 10.Other active autoimmune or inflammatory disorders. 11.Stroke, intracranial haemorrhage, or seizure within 6 months of apheresis. 12.Active uncontrolled epilepsy. 13.Cardiac disease, including arrhythmias, QT prolongation, cardiomyopathy and unstable ischaemic heart disease.

  14.Uncontrolled intercurrent illness. 15.Steroids or other immunomodulators of systemic therapeutic dose within 14 days prior to apheresis.

  16.Prior pegylated G-CSF within 60 days before apheresis. Prior G-CSF/granulocyte-macrophage colony stimulating factor (GM-CSF) within 14 days before apheresis.

  17.Any prohibited medication. 18.Major surgery within 2 weeks prior to apheresis, or planned surgery within 4 weeks after study intervention.

  19.Any history of life-threatening allergies, hypersensitivity, or severe infusion reaction to monoclonal antibodies or biological therapies, or intolerance to the CAR-T product or its excipients.

  20.Toxicity from previous anticancer therapy that has not resolved to baseline levels or to ≤ Grade 1 prior to apheresis.

  21.Female participants who are pregnant or breastfeeding or expect to be pregnant or breastfeeding during the study.

  22.Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

  23.Receipt of live or live attenuated vaccine within 30 days prior to the start of lymphodepletion.

  24.Participant has any medical or psychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs, AESIs, and SAEs. | Within 24 months of the last AZD6422 infusion or the start of a new anticancer treatment
  Incidence of treatment-emergent AEs, AESIs, and SAEs.
Occurrence of Dose limiting toxicity. | Within 28 days after the first infusion
  Occurrence of DLTs (Dose limiting toxicity).
Changes from baseline in vital signs, laboratory parameters, physical examination, and 12-lead ECG. | Within 28 days after the first infusion
  Changes from baseline in vital signs, laboratory parameters, physical examination, and 12-lead ECG.

SECONDARY OUTCOMES:
ORR | 24 months post AZD6422 infusion
  The proportion of participants who have a confirmed CR or confirmed PR as determined by the investigator at local site per RECIST v1.1.
DoR | 24 months post AZD6422 infusion
  The time from first documented confirmed response until date of documented progression of disease per RECIST v1.1 as determined by investigator at local site or death due to any cause.
DCR | 24 months post AZD6422 infusion
  The proportion of participants who have a confirmed CR, confirmed PR, or who have SD per RECIST v1.1 as assessed by the investigator at local site and derived from the raw tumor data for at least 11 weeks after infusion date.
PFS | 24 months post AZD6422 infusion
  Time from infusion date until progression per RECIST v1.1 as assessed by the investigator at local site, or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- peking university Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from sponsor or the collaborator group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the sponsor disclosure commitment. Yes, indicates that sponsors are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: Sponsor or the collaborator group of companies will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to disclosure commitment.
Access Criteria: When a request has been approved sponsor will provide access to the de-identified individual patient-level detain an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
URL: https://vivli.org/